CLINICAL TRIAL: NCT03953430
Title: Normalization of Forefoot Supination After Tibialis Anterior Tendon Transfer for Dynamic Clubfoot Recurrence
Brief Title: Gait Analysis in Children With Clubfoot Treated With Tibialis Anterior Tendon Transfer
Status: Completed | Type: Observational
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Christof Radler, Christof Radler, MD (Head of Pediatric Orthopaedic Team), Orthopedic Hospital Vienna Speising
Other Study IDs: TATT
Record Dates: First submitted 2019-05-03; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Clubfoot
Keywords: Tibialis anterior tendon transfer; Oxford foot model; gait analysis
MeSH Terms: conditions — Clubfoot | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: Patients with clubfoot recurrence undergoing Tibialis Anterior tendon transfer with a minimum age of three years from a prospective, consecutive database of patients with clubfoot treated with the Ponseti method.
  Interventions: Other: Gait analysis
- control group: healthy children of employees of our hospital
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis

SUMMARY:
Patients with clubfoot treated with the Ponseti method and undergoing Tibialis Anterior tendon transfer from a prospective database are evaluated using gait analysis including the Oxford foot model and compared to a group of healthy children.

DETAILED DESCRIPTION:
Children with dynamic clubfoot recurrence after initial Ponseti treatment who underwent TATT between 2014 and 2017 are considered for this study. Exclusion criteria are neurological disease, split transfer of the tendon, additional bone or joint invasive surgery, and initial treatment abroad.

Gait analysis, including the Oxford foot model, will be conducted, and the kinematic and kinetic data of the lower extremity will be compared with a group of age-matched healthy children. To comprise a control group for the purpose of collecting gait analysis data of healthy children, employees of our hospital are asked to allow their children to participate in this study.

Patients will undergo gait analysis, including video recordings with a Vicon motion capture system (Vicon, Oxford, UK) with kinetic data collected from three AMTI force plates (Advanced Mechanical Technology, Inc., Watertown, MA). Placement of markers will be a combination of Cleveland (lower extremity), PlugInGait (upper body), and Oxford Foot (movement within the foot) models.

ELIGIBILITY:
Inclusion Criteria:

* Children with unilateral or bilateral idiopathic clubfoot treated with the Ponseti method
* full TATT

Exclusion Criteria:

* clubfoot associated with syndromes or neurological diseases
* initial Treatment elsewhere with more than 3 casts
* prior joint invasive or bony surgery
* split transfer of the tibialis anterior tendon

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with dynamic clubfoot recurrence with a minimum age of three years from a prospective, consecutive database of patients with clubfoot treated with the Ponseti method
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in forefoot supination in relation to hindfoot after TATT during swing | preoperative (1-21 days) and 6-12 months postoperatively
  The primary outcome measure is forefoot supination in relation to the hindfoot during swing. Changes of forefoot supination during swing after TATT (6-12 months postoperatively) are compared to preoperative values (Oxford foot model). The parameter is a mean value (in degree) of swing phase supination.
  Therefore gait analysis, including video recordings with a Vicon motion capture system (Vicon, Oxford, UK) with kinetic data collected from three AMTI force plates (Advanced Mechanical Technology, Inc., Watertown, MA) will be conducted. Placement of markers will be a combination of Cleveland (lower extremity), PlugInGait (upper body), and Oxford Foot (movement within the foot) models.
  Analysis will include graphic gait curve analysis as well as statistical analysis of pre- to postoperative changes.
Changes in forefoot adduction in relation to hindfoot after TATT during swing | preoperative (1-21 days) and 6-12 months postoperatively
  Another primary outcome measure is forefoot adduction in relation to the hindfoot during swing. Changes of forefoot adduction during swing after TATT (6-12 months postoperatively) are compared to preoperative values (Oxford foot model). The parameter is a mean value (in degree) of swing phase adduction.
  Therefore gait analysis, including video recordings with a Vicon motion capture system (Vicon, Oxford, UK) with kinetic data collected from three AMTI force plates (Advanced Mechanical Technology, Inc., Watertown, MA) will be conducted. Placement of markers will be a combination of Cleveland (lower extremity), PlugInGait (upper body), and Oxford Foot (movement within the foot) models.
  Analysis will include graphic gait curve analysis as well as statistical analysis of pre- to postoperative changes.

CONTACTS AND LOCATIONS:
Overall Officials: Christof Radler, MD, Study Director — Orthopedic Hospital Vienna Speising

REFERENCES:
- [Background] Mindler GT, Kranzl A, Lipkowski CA, Ganger R, Radler C. Results of gait analysis including the Oxford foot model in children with clubfoot treated with the Ponseti method. J Bone Joint Surg Am. 2014 Oct 1;96(19):1593-9. doi: 10.2106/JBJS.M.01603. PMID 25274784